CLINICAL TRIAL: NCT05515107
Title: Inönü University Department of Anesthesia
Brief Title: The Laryngoscopic View With C-MAC Videolaryngoscope Miller Blade Lifting the Epiglottis or the Vallecula in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zekine Begec, Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C-Mac 2
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Intubation; Laryngoscopy
Keywords: Infant; glottis; Laryngoscopy; Intubation

STUDY DESIGN:
Intervention Model Description: Randomized Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blade will placed on vallecula (Active Comparator): Active Comparator: Children will be intubated by the C-MAC VL size 1 Miller blade will placed on the base of the tongue (vallecula)
  Interventions: Device: Videolaryngoscope size 1 Miller blade
- Blade will placed under the epiglottis (Placebo Comparator): Placebo Comparator: Children will be intubated by the C-MAC VL size 1 Miller blade will placed under the epiglottis
  Interventions: Device: Videolaryngoscope size 1 Miller blade

INTERVENTIONS:
Device: Videolaryngoscope size 1 Miller blade — An intubating device that is used for endotracheal intubation. Endotracheal intubation will be performed by anesthesiologist with C-MAC videolaryngoscope

SUMMARY:
In this study, the investigators aim to evaluate the glottic visualization and time to intubation during laryngoscopy performed with the C-MAC VL size 1 Miller blade lifting the epiglottis or placing the tip of the blade on the base of the tongue (vallecula) in children younger than 2 years of age.

DETAILED DESCRIPTION:
Direct laryngoscopy (DL) is the most widely used method to ensure airway safety. In pediatric patients under two years of age, Miller laryngoscope blade is recommended as it removes the long and drooping epiglottis from the eye during laryngoscopy and shows the laryngeal entrance better.

In the classical definition, the tip of the Miller blade is placed behind the epiglottis. However, if the intubator wishes, the Miller blade tip can be placed on the root of the tongue (vallecula) and used as a Macintosh blade.

In the literature search, no study has been found so far comparing C-MAC VL 1 numbered Miller blade with intubation by removing the epiglottis or placing the blade on the vallecula. In this study, the investigators aimed to evaluate the glottic image and intubation time during laryngoscopy performed by lifting the epiglottis with the C-MAC VL No. 1 Miller blade or placing the tip of the blade on the base of the tongue in children under 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 2 years of age
* ASA I and II patients
* Elective surgery under general anesthesia with tracheal intubation

Exclusion Criteria:

* upper respiratory tract infection within the previous 4 weeks
* airway difficulties in the preoperative evaluation
* unstable reactions during intubation

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Percentage of glottic opening score | immediately before endotracheal intubation
  Percentage of glottic opening score of 100% denotes visualization of the entire glottis, from the anterior commissure of the vocal cords to the inter-arytenoid notch. If no part of the glottic opening was visualized, the POGO score was recorded as 0%

SECONDARY OUTCOMES:
Time to intubation | From beginning of holding videolaryngoscope to seeing two meaningful end-tidal carbon dioxide levels up to 3 minutes
  Time to intubation will be measured from the time the videolaryngoscope entered the patient's mouth until the first capnograph trace is seen on the monitor

CONTACTS AND LOCATIONS:
Overall Officials: Zekine Begec, Professor, Study Chair — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Varghese E, Kundu R. Does the Miller blade truly provide a better laryngoscopic view and intubating conditions than the Macintosh blade in small children? Paediatr Anaesth. 2014 Aug;24(8):825-9. doi: 10.1111/pan.12394. Epub 2014 Apr 2. PMID 24690084